CLINICAL TRIAL: NCT05262595
Title: A Study Investigating the Pharmacokinetic and Pharmacodynamic Properties and Safety and Tolerability of Three Formulations of NNC0471-0119 When Administered as One Bolus in a Continuous Subcutaneous Insulin Infusion Regimen in Participants With Type 1 Diabetes
Brief Title: A Study to Look at How Insulin NNC0471-0119 Works in the Body in People With Type 1 Diabetes When Injected by Insulin Pump
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1471-4752; U1111-1260-0359 (Other: World Health Organization (WHO)); 2020-005145-16 (EudraCT Number)
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): A single dose of NNC0471-0119 A, NNC0471-0119 B, NNC0471-0119 D and Faster Aspart at each of 4 visits in random order (four period cross-over)
  Interventions: Drug: NNC0471-0119 A
- Arm 2 (Experimental): A single dose of NNC0471-0119 A, NNC0471-0119 B, NNC0471-0119 D and Faster Aspart at each of 4 visits in random order (four period cross-over)
  Interventions: Drug: NNC0471-0119 B
- Arm 3 (Experimental): A single dose of NNC0471-0119 A, NNC0471-0119 B, NNC0471-0119 D and Faster Aspart at each of 4 visits in random order (four period cross-over)
  Interventions: Drug: NNC0471-0119 D
- Arm 4 (Active Comparator): A single dose of NNC0471-0119 A, NNC0471-0119 B, NNC0471-0119 D and Faster Aspart at each of 4 visits in random order (four period cross-over)
  Interventions: Drug: Faster aspart

INTERVENTIONS:
Drug: NNC0471-0119 A — NNC0471-0119 administered once via an insulin pump as one bolus dose on top of a continuous basal rate.
  The study will last 1-4 months
  Arms: Arm 1
Drug: NNC0471-0119 B — NNC0471-0119 administered once via an insulin pump as one bolus dose on top of a continuous basal rate.
  The study will last 1-4 months
  Arms: Arm 2
Drug: NNC0471-0119 D — NNC0471-0119 administered once via an insulin pump as one bolus dose on top of a continuous basal rate.
  The study will last 1-4 months
  Arms: Arm 3
Drug: Faster aspart — Faster aspart administered once via an insulin pump as one bolus dose on top of a continuous basal rate.
  The study will last 1-4 months
  Arms: Arm 4

SUMMARY:
This study is looking at the effect and safety of 3 formulations of the new rapid-acting insulin analogue NNC0471-0119, for the treatment of type 1 diabetes when given by insulin pump.

The study will test how 3 different formulations of insulin NNC0471-0119 are tolerated by the body, how they are transported in participants bloodstream, how long they stay there and how the blood sugar is lowered.

The 3 formulations of insulin NNC0471-0119 are given as one bolus on top of a constant insulin basal rate and compared to Faster Aspart (Fiasp®).

Participants will get 3 formulations of insulin NNC0471-0119 and Faster Aspart (Fiasp®) Insulin NNC0471-0119 is a new rapid-acting insulin designed to be used in an insulin pump. Faster Aspart (Fiasp®) is a globally used medication for the treatment of diabetes.

Participants will have each study medicine administered once via pump at separate study visits. This mean that participants will have a total of 4 dosing visits where participants will get a study medicine. Which study medicine participants get at what visit will be decided by chance.

The study will last 1-4 months. Participants will have 7 visits at the clinic, 4 of them will require an in-house stay of 3 consecutive days each.

During the in-house visits 2 intravenous (into the vein) cannulas will be inserted for blood sampling and infusions.

Women: Women cannot take part if they are of childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Male participant or female participant of non-childbearing potential. Non-childbearing potential being defined as surgically sterilised (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy) or being postmenopausal (defined as no menses for 12 months without an alternative medical cause) prior to the day of screening.
* Aged 18-64 years (both inclusive) at the time of signing informed consent.
* Diagnosed with T1DM for more than1 year prior to the day of screening.
* Current total daily insulin treatment between 0.2 and 1.2 (I)U/kg/day (both inclusive).
* Treated with continuous subcutaneous insulin infusion greater than 90 days prior to the day of screening.

Exclusion Criteria:

* Known or suspected hypersensitivity to study interventions or related products.
* Participation (i.e., study intervention) in any interventional, clinical study within 30 days or 5 times the half-life of the drug, whichever is longest before screening.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
AUC (NNC0471-0119,0-30min,basal-corrected)/AUC (NNC0471-0119,0-t,basal-corrected) | 0 to 12 hours after bolus infusion
  Ratio of the basal-corrected area under the serum NNC0471-0119 concentration time curve from 0 to 30 minutes and 0 to t, where t is the first time the curve is back to basal level after bolus infusion (at most 12 hours).
  Measured in percentage

SECONDARY OUTCOMES:
AUC (NNC0471-0119,0-t,basal-corrected) | 0 to 12 hours after bolus infusion
  Area under the basal-corrected serum NNC0471-0119 concentration time curve from 0 to t, where t is the first time the curve is back to basal level after bolus infusion (at most 12 hours).
  Measured in h*pmol/L
AUC (NNC0471-0119,0-30min,basal-corrected) | 0 to 30 minutes after bolus infusion
  Area under the basal-corrected serum NNC0471-0119 concentration time curve from 0 to 30 minutes.
  Measured in h*pmol/L
AUC (NNC0471-0119,2h-t,basal-corrected) | 2 to 12 hours after bolus infusion
  Area under the basal-corrected serum NNC0471-0119 concentration time curve from 2 hours to t, where t is the first time the curve is back to basal level after bolus infusion (at most 12 hours).
  Measured in h*pmol/L
AUC (NNC0471-0119,2h-t,basal-corrected)/AUC (NNC0471-0119,0-t,basal-corrected) | 0 to 12 hours after bolus infusion
  Ratio of the basal-corrected area under the serum NNC0471-0119 concentration time curve from 2 hours to t and 0 to t, where t is the first time the curve is back to basal level after bolus infusion (at most 12 hours).
  Measured in percentage
Cmax,NNC0471-0119,basal-corrected: Maximum observed basal-corrected serum NNC0471-0119 concentration | 0 to 12 hours after bolus infusion
  pmol/L
Number of adverse events (AEs) | From start of first investigational medicinal product ( IMP) basal rate infusion (Visit 2, day -1) until completion of post-treatment end-of-study visit (Visit 6)
  Number of events
AUC (GIR,0-t,basal-corrected) | 0 to 12 hours after bolus infusion
  Area under the basal-corrected glucose infusion rate (GIR)-time curve from 0 to t, where t is the first time the GIR curve is back to basal level after bolus infusion (at most 12 hours).
  Measured in mg/kg
AUC (GIR,0-1h,basal-corrected) | 0 to 1 hour after bolus infusion
  Area under the basal-corrected GIR-time curve from 0 to 1 hour. Measured in mg/kg
AUC (GIR,0-1h,basal-corrected/AUC (GIR,0-t,basal-corrected) | 0 to 12 hours after bolus infusion
  Ratio of the area under the basal-corrected GIR-time curve from 0 to 1 hour and 0 to t, where t is the first time the GIR curve is back to basal level after bolus infusion (at most 12 hours).
  Measured in percentage
GIRmax,basal-corrected: Maximum observed basal-corrected GIR | 0 to 12 hours after bolus infusion
  mg/(kg*min)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com